CLINICAL TRIAL: NCT03091231
Title: Multiparametric Ultrasound - Contrast Enhanced Ultrasound and Shear Wave Elastography Compared to Radical Prostatectomy Specimens in 50 Patients
Brief Title: Multiparametric Ultrasound-Study for the Detection of Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Martini-Klinik am UKE GmbH (Other)
Collaborators: Eindhoven University of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: mpUS-Study_2016
Record Dates: First submitted 2017-03-14; First posted 2017-03-27 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: mpUS multiparametric Ultrasound — compare the mpUS to other methods

SUMMARY:
The primary objective of the study is the matching of sensitivity, specificity, the negative predicate value and the positive predictive value of Contrast-Enhanced Ultrasound (CEUS), Shear Wave Elastography (SWE) and the combination to detect clinically significant prostate carcinoma foki.

Conventional ultrasound is insufficient to safely display prostate carcinoma. Therefore, other imaging agents are recently added to improve the detection of tumor foci. These include innovative imaging ultrasound methods and multiparametric MRI.

DETAILED DESCRIPTION:
All patients scheduled for radical prostatectomy in the Martini-Klinik are admitted the day prior to the surgery. In case a patient gives his informed consent mpUS (multiparametric Ultrasound) scanning is performed on the day prior to surgery, the day of admittance. The patient will be prepared with an intravenous access to administer the contrast agent. Ultrasound Scanning will be performed in the left-lateral decubitus position and start with regular B-mode scanning and volumetry. A base to apex sweeps and left to right sweep will be acquired to allow building a 3D reconstruction of the prostate. The imaging protocol will then start with SWE. Stiffness of the tissue is measured in Shear modulus (kPa) and visualized in a color scale. SWE results will be recorded for later interpretation and analysis. Then 2 minute recordings of CEUS imaging will be made following the administration of a 2.4ml bolus of the contrast agent SonoVue® (Bracco, Geneva) through the intravenous canula. A maximum of four recordings will be made. For every recording a new bolus of contrast agent will be administered. In this way, for planes the contrast inflow can be recorded. Data will be stored and transported to an image processing system for dispersion analysis. On this system a dispersion (CUDI) parametric map will be constructed from each acquired CEUS recording. At the time of interpretation imaging results will be scored separately for the standard prostate sextants, base left, base right, mid left, mid right, apex left and apex right.

The radical prostatectomy will be performed as in accordance to institution standards. This procedure will not be altered because of the trial. In many cases this means frozen sections are taken intraoperatively from the lateral sides of the prostate. These frozen sections are processed separately from the resection specimen in the pathology lab. Following the radical prostatectomy the resection specimen is fixated according to institution standards. This means that the specimen is photographed and the location and orientation of all coupes is recorded. This will enable allocating pathology findings to the standard prostate sextants described earlier.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* signed informed consent

Exclusion Criteria:

* History of any clinically evidence of cardiac right-to-left shunts
* Receives treatment that includes dobutamine
* Severe pulmonary hypertension (pulmonary artery pressure >90 mmHg) or uncontrolled systemic hypertension or respiratory distress syndrome
* Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study
* Is incapable of understanding the language in which the information for the patient is given

Ages: 18 Years to 75 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — only men get prostate cancer
Study Population: All patients scheduled for radical prostatectomy in the Martini Klinik that fulfil the inclusion criteria and do not have any of the exclusion criteria are eligible for participation in this study. Patients will be informed about the objectives, procedures and risks of the study all patients will have to sign written informed consent prior to participation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy in terms of sensitivity and specificity of CEUS, SWE and their combination using radical prostatectomy specimens as the gold-standard. | 14 days
  The data gathered will be structured so that for each prostate sextant B-mode TRUS results, SWE results, CEUS results including CUDI maps and Pathology results are available for correlation. For the imaging modalities quantifiable data and visual interpretation using a 1 to 5 Likert-type scale for suspicion will be stored for each sextant. Pathology data will be gathered in the form of tumor size and grade. The data will be used to calculate sensitivity, specificity, negative predictive value and positive predictive value for each of the imaging modalities separately. Furthermore the data will be used to calculate an optimal algorithm for combining the imaging modalities. The maximum attainable sensitivity, specificity, NPV and PPV for tumor detection using this optimized algorithm will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Georg Salomon, PD Dr., Principal Investigator — Martini-Klinik am UKE GmbH
Locations (1):
- Martini-Klinik am UKE GmbH, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
Anonymized data from ultrasound results and histological findings are sent to the TU Eindhoven in Eindhoven (Netherlands) for quantification analysis.

REFERENCES:
- [Derived] Mannaerts CK, Wildeboer RR, Postema AW, Hagemann J, Budaus L, Tilki D, Mischi M, Wijkstra H, Salomon G. Multiparametric ultrasound: evaluation of greyscale, shear wave elastography and contrast-enhanced ultrasound for prostate cancer detection and localization in correlation to radical prostatectomy specimens. BMC Urol. 2018 Nov 8;18(1):98. doi: 10.1186/s12894-018-0409-5. PMID 30409150
- Available data/document: Study Protocol: mpUS2016 — http://www.martini-klinik.de — to request an electronic copy send an email to a.renter@uke.de